CLINICAL TRIAL: NCT00665795
Title: Morphometric Analysis of Orbital Structures in Graves´ Orbitopathy Using Multidetector Computed Tomography Scan and Color Doppler Imaging.
Brief Title: Morphometric Analysis of Orbital Structures in Graves´ Orbitopathy
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Allan Christian Pieroni Goncalves, MD, University of Sao Paulo
Other Study IDs: 1152/05
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Dysthyroid Orbitopathy
Keywords: Dysthyroid Optic Neuropathy; multidetector computed tomography; color doppler; Grave´s Orbitopathy; Grave´s Disease; morphometric analysis
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1Patients with Graves´orbitophathy.: Patients with Graves´orbitophathy.
- 2 Patients with detected DON: Patients with Graves´orbitophaty and detected dysthyroid optic neuropathy (DON)

SUMMARY:
The purpose of this protocol is to study orbital structures in Graves´ Disease using multidetector computed tomography and color doppler imaging.

Some changes in orbital structures detected by imaging exams could predict severity of the ocular Graves´disease. Thus the study could be useful in improve medical management of patients with Graves´ Disease.

DETAILED DESCRIPTION:
Morphometric analysis of orbital structures in Graves´ Orbitopathy using multidetector computed tomography scan and color doppler imaging:

Patients with Graves´ orbitopathy are evaluated by a complete ophthalmic examination.A prospective study with Multidetector CT scan and Color Doppler of these patients are made to develop parameters capable to predict Dysthyroid Optic Neuropathy (DON).

ELIGIBILITY:
Inclusion Criteria:

* Graves´Orbitopathy diagnosed based on previously reported criteria
* Age above 20 years
* Good cooperation for performing Visual Field test
* Spherical refraction within ± 5 D and cylinder correction within ± 3 D

Exclusion Criteria:

* Graves´Orbitopathy not diagnosed

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Graves´ orbitopathy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2005-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
screening indexes for dysthyroid optic neuropathy | indexes above 60% of orbital apex crowding were high suspected for DON

CONTACTS AND LOCATIONS:
Overall Officials: Mario L Monteiro, MD, PhD, Study Chair — University of Sao Paulo - School of Medicine
Locations (1):
- General Hospital - University of Sao Paulo - School of Medicine, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Goncalves AC, Silva LN, Gebrim EM, Monteiro ML. Quantification of orbital apex crowding for screening of dysthyroid optic neuropathy using multidetector CT. AJNR Am J Neuroradiol. 2012 Sep;33(8):1602-7. doi: 10.3174/ajnr.A3029. Epub 2012 Mar 22. PMID 22442048